CLINICAL TRIAL: NCT00462436
Title: Do Innovative Strategies Complement Medical Management to Reduce Cardiovascular Risk Factors Following Coronary Artery Bypass Graft Surgery?
Brief Title: Innovative Strategies For Risk Reduction Following CABG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Dr. Mary Keith, St. Michael's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB06-179C
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Disease; Type II Diabetes Mellitus
Keywords: functional foods; soy; nuts; LDL cholesterol; fibre; secondary prevention; risk reduction; endothelial function; endothelial progenitor cells; inflammation; glycemic control; HOMA
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Risk Reduction Behavior; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Consumption of Dietary Portfolio — The study involves following an aggressive low fat diet that is high in viscous fiber, nuts and soy protein. The diet is individually tailored to meet individual participants needs.

SUMMARY:
Background: Treatment targets for cardiac risk factor reduction are not being met. Therefore, there is a need for new strategies to assist patients in meeting these goals.

Objective: To determine the amount of any additional benefit on risk factor reduction associated with the consumption of the "dietary portfolio" (a low fat diet with soy, nuts and viscous fibres), above that achieved with medical management in diabetic patients following cardiac surgery.

Description: 35 cardiac surgery patients with diabetes will be instructed on how to incorporate the dietary portfolio foods into their diet for four weeks. Changes in blood cholesterol, markers of inflammation, blood sugar control and modifiable risk factors will be assessed after 2 and 4 weeks of therapy.

Relevance: Maximizing cardiac risk factor reduction through a combined approach (dietary plus medication) should improve outcomes, reduce rates of re-hospitalization and improve quality of life in diabetic patients after heart surgery.

DETAILED DESCRIPTION:
Introduction: The consumption of a dietary portfolio has been found to successfully reduce LDL cholesterol by 30% in hyperlipidemic, non-diabetic patients under highly controlled conditions. Given the burden of cardiovascular disease in the diabetic population, it is now important that we evaluate whether consumption of the dietary portfolio can reduce modifiable risk factors and improve diabetic control above that associated with medical therapy alone in this population. The reduction of modifiable risk factors, particularly in the diabetic patient with coronary artery disease, should not only improve long-term outcomes thereby reducing re-admissions and subsequently the burden of the diabetic patient on the health care system, but also improve quality of life for these patients. This pilot project will determine the efficacy, feasibility and tolerability of an aggressive dietary strategy, the dietary portfolio of functional foods to reduce cardiovascular risk factors in diabetic patients following CABG.

Study Objectives: This study will determine to what extent the self selected "modified" dietary portfolio (without sterols) together with statin therapy will:

* reduce total and LDL cholesterol
* increase endothelial cell number and function and reduce CRP levels.
* reduce markers of inflammation and insulin resistance
* the study will also determine the tolerability of and compliance with the portfolio diet

Primary Hypothesis: The consumption of the modified dietary portfolio will have a pleiotropic effect with current statin therapy resulting in an additional reduction in LDL cholesterol of 25% after four weeks of treatment.

Secondary Hypotheses: The addition of the dietary portfolio together with statin therapy will:

* significantly increase measures of endothelial function and endothelial progenitor cell counts
* significantly reduce CRP levels
* be feasible and well tolerated by most bypass patients
* result in a compliance rate of 70% with the main components of the diet
* significantly improve the plasma total-C:HDL-C ratio, and total-C, HDL-C, apolipoproteins A-I and B levels after both two and four weeks of treatment
* significantly reduce markers of inflammation at four weeks (CRP, IL-6 and TNF)
* improve indices of glycemic control (HOMA), oxidized LDL and LDL particle size

Trial Design:

Subject Selection: Participants will be screened from those patients returning for their routine six week follow-up visit following their coronary artery bypass graft surgery. Eligible patients will be invited to participate in this secondary prevention trial by their surgeon. The six week time point for recruitment not only allows direct patient interaction but also ensures that sufficient time has passed for normalization of the lipid profile post CABG (20). Finally, at this time, most patients have also seen their cardiologist and have had their medication regimen adjusted following surgery, which should allow for a window of stable medical care over the course of the study.

Patients with type II diabetes are selected for this study as 1) this group of patients is at a higher risk of developing post-operative complications and therefore are most likely to receive the maximal benefit from risk factor modification, and 2) this group has increased cardiovascular risk and therefore should benefit on multiple levels by the addition of the portfolio diet including, but not limited to reduced LDL cholesterol, blood pressure, CRP and inflammatory response but also in improved insulin sensitivity and endothelial function. Finally since estrogen levels influence endothelial function, pre-menopausal women will be excluded from this pilot study.

Study Design: This is non-randomized pilot study investigating the magnitude of cardiovascular risk reduction achieved by the addition of a "modified portfolio diet" (DPF)(without plant sterols) consumed for one month under real life conditions in diabetic patients on statin therapy who have known cardiovascular disease. The four week intervention period has previously been found to be sufficient for significant changes in the primary outcome variable (LDL cholesterol) to occur but will be short enough to minimize the confounding effects of changes in medication and physical activity in hypercholesterolemic subjects not on statin therapy(21).

The study will involve one baseline and two follow-up visits (Figure 1). At baseline, demographic, anthropometric (weight, height, body mass index (BMI), waist/hip ratio) and medical/cardiac history will be obtained including a detailed list of current medications. Resting blood pressure will be measured (see analytic methods). Information regarding exercise and smoking habits will also be obtained at this time. Participants will receive comprehensive dietary advice by a trained registered dietitian at the Risk Factor Modification Centre. The DPF group will conform to current therapeutic diets appropriate for hypercholesterolemic subjects (<7% of energy saturated fat, <200 mg/d cholesterol) with the addition of a combination of viscous fibers, soy protein and almonds. Participants will be instructed on how to select and follow this diet and will be provided with samples of appropriate foods to assist in the initial selection of and compliance with the DPF. All participants will receive a weekly allowance for the purchase of appropriate foods. The portfolio diet plan will include foods which contribute 8 g/1000 kcal viscous fiber as β-glucan (oats, barley, oat bran breads and soups) and psyllium (cereal), 17 g soy protein/1000 kcal (soy burgers, hot dogs, links, other meat analogues, milks, yogurts and cheese) and 22 g nuts (almonds)/1000 kcal. Participants at the Risk Factor Modification Centre have been maintained on this level of fiber intake for 4-month periods (22). Moderate weight loss (0.5kg/week) for those with a BMI >25 and routine physical activity using the guidelines from the Guide to Cardiac surgery will be encouraged as part of this secondary prevention strategy. During the baseline visit, the coordinator (MSc student) will complete a 24 hour dietary recall to obtain an idea of estimated dietary intake. This recall together with calculated energy requirements using established equations will be used to assess individual energy intake. Using this estimate, the coordinator will advise the participant on how to incorporate the DPF into their eating patterns. The coordinator will instruct patients on detailed diet history recording, and each participant will be provided printed booklets in which to record the food items and their approximate size. Since determining compliance is an important end-point, self-taring scales will be provided to assist with accuracy. Subjects will be asked to complete daily a checklist of their consumption of the three key foods or food components of the portfolio diet (23,24). Assessment of the checklists for the three key dietary components will provide not only an estimate of compliance but will also assist patients in monitoring on a daily basis how many foods from the portfolio they have consumed. The coordinator will complete 4 random 24 hour recalls with each study subject, using standardized techniques, throughout the study period in order to validate the compliance checklist data. Recall data will be analyzed using a program based on USDA data (25) with additional data on foods analyzed in the laboratory for protein, total fat, and dietary fiber using the methods of the Association of Official Analytical Chemists (AOAC) (26) as well as the tables of Anderson and Bridges (27).

Since the DPF is part of a comprehensive secondary prevention strategy, all participants will be encouraged to follow the guidelines for physical activity (30 minutes, 3-5 times per week) outlined in the Guide for Cardiac Surgery Outpatient Handbook. The amount of physical activity will be recorded using a pedometer and will be recorded at the bottom of their food checklist. Fasting blood samples will be collected for primary and secondary markers of cardiovascular risk, insulin resistance and endothelial function. Brachial artery vasoreactivity will be completed at the same time of day with each participant under fasting conditions. Medications will be held the morning of the test.

Significance of Proposal: This study will determine the magnitude of any additional cardiovascular risk reduction associated with the consumption of the "modified dietary portfolio" in diabetic patients with coronary artery disease on statin therapy. Furthermore, since the dietary portfolio is an aggressive strategy, this study will also determine the feasibility and tolerability of this type of intervention in patients living in the community. Finally, this study may justify a larger secondary prevention trial looking at the effect of this intervention on cardiac outcomes and rates of re-hospitalization following bypass grafting. Aggressive, innovative, patient driven dietary strategies may complement medical management improving the ability of patients to meet treatment targets ultimately resulting in improved patient outcomes and quality of life following bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type II diabetes mellitus
2. Recently (<5 months) undergone coronary artery bypass graft surgery
3. Taking cholesterol lowering medication

Exclusion Criteria:

1. Can not speak English and have no available interpreter
2. Refuse Informed Consent
3. Had "off pump" CABG
4. Are intolerant of statins
5. Are pre-menopausal (women) or are on HRT
6. Have serious concomitant disease
7. Take insulin
8. Are <18 years of age
9. receive incomplete revascularization
10. documented history of drug or alcohol abuse
11. Intend to become pregnant during study period
12. Have an unreliable psychological condition that makes them unlikely to comply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Reduction of total and LDL cholesterol | baseline to 4 weeks

SECONDARY OUTCOMES:
Improvement in endothelial function and EPC counts | Baseline to 4 weeks
Reduction in CRP | baseline to 4 weeks
Feasibility and tolerability | Baseline to 4 Weeks
Reduction in markers of inflammation ie TNF, IL-6 | Baseline to 4 weeks
Improved markers of glycemic control - fructosamine, HOMA | baseline to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary Keith, PhD, RD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Herlitz J, Wognsen GB, Emanuelsson H, Haglid M, Karlson BW, Karlsson T, Albertsson P, Westberg S. Mortality and morbidity in diabetic and nondiabetic patients during a 2-year period after coronary artery bypass grafting. Diabetes Care. 1996 Jul;19(7):698-703. doi: 10.2337/diacare.19.7.698. PMID 8799622
- [Background] Morricone L, Ranucci M, Denti S, Cazzaniga A, Isgro G, Enrini R, Caviezel F. Diabetes and complications after cardiac surgery: comparison with a non-diabetic population. Acta Diabetol. 1999 Jun;36(1-2):77-84. doi: 10.1007/s005920050149. PMID 10436257
- [Background] Carson JL, Scholz PM, Chen AY, Peterson ED, Gold J, Schneider SH. Diabetes mellitus increases short-term mortality and morbidity in patients undergoing coronary artery bypass graft surgery. J Am Coll Cardiol. 2002 Aug 7;40(3):418-23. doi: 10.1016/s0735-1097(02)01969-1. PMID 12142105
- [Background] Schwartz L, Kip KE, Frye RL, Alderman EL, Schaff HV, Detre KM; Bypass Angioplasty Revascularization Investigation. Coronary bypass graft patency in patients with diabetes in the Bypass Angioplasty Revascularization Investigation (BARI). Circulation. 2002 Nov 19;106(21):2652-8. doi: 10.1161/01.cir.0000038885.94771.43. PMID 12438289
- [Background] Post Coronary Artery Bypass Graft Trial Investigators. The effect of aggressive lowering of low-density lipoprotein cholesterol levels and low-dose anticoagulation on obstructive changes in saphenous-vein coronary-artery bypass grafts. N Engl J Med. 1997 Jan 16;336(3):153-62. doi: 10.1056/NEJM199701163360301. PMID 8992351
- [Background] Pearson TA, Peters TD. The treatment gap in coronary artery disease and heart failure: community standards and the post-discharge patient. Am J Cardiol. 1997 Oct 30;80(8B):45H-52H. doi: 10.1016/s0002-9149(97)00820-5. PMID 9372998
- [Background] EUROASPIRE I and II Group; European Action on Secondary Prevention by Intervention to Reduce Events. Clinical reality of coronary prevention guidelines: a comparison of EUROASPIRE I and II in nine countries. EUROASPIRE I and II Group. European Action on Secondary Prevention by Intervention to Reduce Events. Lancet. 2001 Mar 31;357(9261):995-1001. doi: 10.1016/s0140-6736(00)04235-5. PMID 11293642
- [Background] Grundy SM, Balady GJ, Criqui MH, Fletcher G, Greenland P, Hiratzka LF, Houston-Miller N, Kris-Etherton P, Krumholz HM, LaRosa J, Ockene IS, Pearson TA, Reed J, Washington R, Smith SC Jr. Primary prevention of coronary heart disease: guidance from Framingham: a statement for healthcare professionals from the AHA Task Force on Risk Reduction. American Heart Association. Circulation. 1998 May 12;97(18):1876-87. doi: 10.1161/01.cir.97.18.1876. No abstract available. PMID 9603549
- [Background] McFarlane SI, Jacober SJ, Winer N, Kaur J, Castro JP, Wui MA, Gliwa A, Von Gizycki H, Sowers JR. Control of cardiovascular risk factors in patients with diabetes and hypertension at urban academic medical centers. Diabetes Care. 2002 Apr;25(4):718-23. doi: 10.2337/diacare.25.4.718. PMID 11919131
- [Background] George PB, Tobin KJ, Corpus RA, Devlin WH, O'Neill WW. Treatment of cardiac risk factors in diabetic patients: How well do we follow the guidelines? Am Heart J. 2001 Nov;142(5):857-63. doi: 10.1067/mhj.2001.119132. PMID 11685175
- [Background] Hiss RG, Anderson RM, Hess GE, Stepien CJ, Davis WK. Community diabetes care. A 10-year perspective. Diabetes Care. 1994 Oct;17(10):1124-34. doi: 10.2337/diacare.17.10.1124. PMID 7821131
- [Background] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; National Heart, Lung, and Blood Institute; American College of Cardiology Foundation; American Heart Association. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III guidelines. Circulation. 2004 Jul 13;110(2):227-39. doi: 10.1161/01.CIR.0000133317.49796.0E. PMID 15249516
- [Background] Ridker PM. Clinical application of C-reactive protein for cardiovascular disease detection and prevention. Circulation. 2003 Jan 28;107(3):363-9. doi: 10.1161/01.cir.0000053730.47739.3c. No abstract available. PMID 12551853
- [Background] Ooi M, Cooper A, Lloyd G, Jackson G. A study of lipid profile before and after coronary artery bypass grafting. Br J Clin Pract. 1996 Dec;50(8):433-5. PMID 9039713
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Lapsley KG, Trautwein EA, Josse RG, Leiter LA, Connelly PW. Effects of a dietary portfolio of cholesterol-lowering foods vs lovastatin on serum lipids and C-reactive protein. JAMA. 2003 Jul 23;290(4):502-10. doi: 10.1001/jama.290.4.502. PMID 12876093
- [Background] Jenkins DJ, Wolever TM, Rao AV, Hegele RA, Mitchell SJ, Ransom TP, Boctor DL, Spadafora PJ, Jenkins AL, Mehling C, et al. Effect on blood lipids of very high intakes of fiber in diets low in saturated fat and cholesterol. N Engl J Med. 1993 Jul 1;329(1):21-6. doi: 10.1056/NEJM199307013290104. PMID 8389421
- [Background] Bingham SA, Gill C, Welch A, Day K, Cassidy A, Khaw KT, Sneyd MJ, Key TJ, Roe L, Day NE. Comparison of dietary assessment methods in nutritional epidemiology: weighed records v. 24 h recalls, food-frequency questionnaires and estimated-diet records. Br J Nutr. 1994 Oct;72(4):619-43. doi: 10.1079/bjn19940064. PMID 7986792
- [Background] Goldberg GR, Black AE, Jebb SA, Cole TJ, Murgatroyd PR, Coward WA, Prentice AM. Critical evaluation of energy intake data using fundamental principles of energy physiology: 1. Derivation of cut-off limits to identify under-recording. Eur J Clin Nutr. 1991 Dec;45(12):569-81. PMID 1810719
- [Background] 25. The Agricultural Research Service. Composition of Foods, Agriculture Handbook No 8. Washington, DC, US Department of Agriculture, 1992.
- [Background] 26. Association of Official Analytical Chemists. AOAC Official Methods of Analysis. Washington, DC, Association of Official Analytical Chemists, 1980.
- [Background] Anderson JW, Bridges SR. Dietary fiber content of selected foods. Am J Clin Nutr. 1988 Mar;47(3):440-7. doi: 10.1093/ajcn/47.3.440. PMID 2831703
- [Background] Fagerberg B, Hulthe J, Bokemark L, Wikstrand J. Low-density lipoprotein particle size, insulin resistance, and proinsulin in a population sample of 58-year-old men. Metabolism. 2001 Jan;50(1):120-4. doi: 10.1053/meta.2001.18570. PMID 11172485
- [Background] Garvey WT, Kwon S, Zheng D, Shaughnessy S, Wallace P, Hutto A, Pugh K, Jenkins AJ, Klein RL, Liao Y. Effects of insulin resistance and type 2 diabetes on lipoprotein subclass particle size and concentration determined by nuclear magnetic resonance. Diabetes. 2003 Feb;52(2):453-62. doi: 10.2337/diabetes.52.2.453. PMID 12540621
- [Background] Lamarche B, St-Pierre AC, Ruel IL, Cantin B, Dagenais GR, Despres JP. A prospective, population-based study of low density lipoprotein particle size as a risk factor for ischemic heart disease in men. Can J Cardiol. 2001 Aug;17(8):859-65. PMID 11521128
- [Background] St-Pierre AC, Ruel IL, Cantin B, Dagenais GR, Bernard PM, Despres JP, Lamarche B. Comparison of various electrophoretic characteristics of LDL particles and their relationship to the risk of ischemic heart disease. Circulation. 2001 Nov 6;104(19):2295-9. doi: 10.1161/hc4401.098490. PMID 11696468
- [Background] Krauss RM. Dense low density lipoproteins and coronary artery disease. Am J Cardiol. 1995 Feb 23;75(6):53B-57B. doi: 10.1016/0002-9149(95)80012-h. PMID 7863975
- [Background] Williams PT, Haskell WL, Vranizan KM, Krauss RM. The associations of high-density lipoprotein subclasses with insulin and glucose levels, physical activity, resting heart rate, and regional adiposity in men with coronary artery disease: the Stanford Coronary Risk Intervention Project baseline survey. Metabolism. 1995 Jan;44(1):106-14. doi: 10.1016/0026-0495(95)90296-1. PMID 7854154
- [Background] Berneis KK, Krauss RM. Metabolic origins and clinical significance of LDL heterogeneity. J Lipid Res. 2002 Sep;43(9):1363-79. doi: 10.1194/jlr.r200004-jlr200. PMID 12235168
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Asahara T, Masuda H, Takahashi T, Kalka C, Pastore C, Silver M, Kearne M, Magner M, Isner JM. Bone marrow origin of endothelial progenitor cells responsible for postnatal vasculogenesis in physiological and pathological neovascularization. Circ Res. 1999 Aug 6;85(3):221-8. doi: 10.1161/01.res.85.3.221. PMID 10436164
- [Background] Takahashi T, Kalka C, Masuda H, Chen D, Silver M, Kearney M, Magner M, Isner JM, Asahara T. Ischemia- and cytokine-induced mobilization of bone marrow-derived endothelial progenitor cells for neovascularization. Nat Med. 1999 Apr;5(4):434-8. doi: 10.1038/7434. PMID 10202935
- [Background] Vasa M, Fichtlscherer S, Aicher A, Adler K, Urbich C, Martin H, Zeiher AM, Dimmeler S. Number and migratory activity of circulating endothelial progenitor cells inversely correlate with risk factors for coronary artery disease. Circ Res. 2001 Jul 6;89(1):E1-7. doi: 10.1161/hh1301.093953. PMID 11440984
- [Background] Tepper OM, Galiano RD, Capla JM, Kalka C, Gagne PJ, Jacobowitz GR, Levine JP, Gurtner GC. Human endothelial progenitor cells from type II diabetics exhibit impaired proliferation, adhesion, and incorporation into vascular structures. Circulation. 2002 Nov 26;106(22):2781-6. doi: 10.1161/01.cir.0000039526.42991.93. PMID 12451003
- [Background] Schachinger V, Britten MB, Zeiher AM. Prognostic impact of coronary vasodilator dysfunction on adverse long-term outcome of coronary heart disease. Circulation. 2000 Apr 25;101(16):1899-906. doi: 10.1161/01.cir.101.16.1899. PMID 10779454
- [Background] Anderson TJ, Uehata A, Gerhard MD, Meredith IT, Knab S, Delagrange D, Lieberman EH, Ganz P, Creager MA, Yeung AC, et al. Close relation of endothelial function in the human coronary and peripheral circulations. J Am Coll Cardiol. 1995 Nov 1;26(5):1235-41. doi: 10.1016/0735-1097(95)00327-4. PMID 7594037
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Verma S, Kuliszewski MA, Li SH, Szmitko PE, Zucco L, Wang CH, Badiwala MV, Mickle DA, Weisel RD, Fedak PW, Stewart DJ, Kutryk MJ. C-reactive protein attenuates endothelial progenitor cell survival, differentiation, and function: further evidence of a mechanistic link between C-reactive protein and cardiovascular disease. Circulation. 2004 May 4;109(17):2058-67. doi: 10.1161/01.CIR.0000127577.63323.24. Epub 2004 Apr 12. PMID 15078802
- [Background] Lieberman EH, Gerhard MD, Uehata A, Selwyn AP, Ganz P, Yeung AC, Creager MA. Flow-induced vasodilation of the human brachial artery is impaired in patients <40 years of age with coronary artery disease. Am J Cardiol. 1996 Dec 1;78(11):1210-4. doi: 10.1016/s0002-9149(96)00597-8. PMID 8960576
- [Background] Jenkins DJ, Kendall CW, Marchie A, Parker TL, Connelly PW, Qian W, Haight JS, Faulkner D, Vidgen E, Lapsley KG, Spiller GA. Dose response of almonds on coronary heart disease risk factors: blood lipids, oxidized low-density lipoproteins, lipoprotein(a), homocysteine, and pulmonary nitric oxide: a randomized, controlled, crossover trial. Circulation. 2002 Sep 10;106(11):1327-32. doi: 10.1161/01.cir.0000028421.91733.20. PMID 12221048
- [Background] Jenkins DJ, Kendall CW, Jackson CJ, Connelly PW, Parker T, Faulkner D, Vidgen E, Cunnane SC, Leiter LA, Josse RG. Effects of high- and low-isoflavone soyfoods on blood lipids, oxidized LDL, homocysteine, and blood pressure in hyperlipidemic men and women. Am J Clin Nutr. 2002 Aug;76(2):365-72. doi: 10.1093/ajcn/76.2.365. PMID 12145008
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Martini MC, Axelsen M, Faulkner D, Vidgen E, Parker T, Lau H, Connelly PW, Teitel J, Singer W, Vandenbroucke AC, Leiter LA, Josse RG. Effect of wheat bran on glycemic control and risk factors for cardiovascular disease in type 2 diabetes. Diabetes Care. 2002 Sep;25(9):1522-8. doi: 10.2337/diacare.25.9.1522. PMID 12196421
- [Derived] Keith M, Kuliszewski MA, Liao C, Peeva V, Ahmed M, Tran S, Sorokin K, Jenkins DJ, Errett L, Leong-Poi H. A modified portfolio diet complements medical management to reduce cardiovascular risk factors in diabetic patients with coronary artery disease. Clin Nutr. 2015 Jun;34(3):541-8. doi: 10.1016/j.clnu.2014.06.010. Epub 2014 Jun 28. PMID 25023926